CLINICAL TRIAL: NCT05688605
Title: An Open-label, Multi-center, Phase I/II Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of MRG003 in Combination With HX008 in Patients With EGFR-positive Advanced Solid Tumors
Brief Title: A Study of MRG003 in the Treatment of Patients With EGFR-positive Advanced or Metastatic Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Miracogen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX008/MRG003-C001
Record Dates: First submitted 2023-01-06; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Advanced Solid Tumors
Keywords: MRG003; HX008; Antibody Drug Conjugate (ADC); EGFR; Solid tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRG003+HX008 (Experimental): MRG003 will be administrated via intravenous infusion at 1.5, 2.0 mg/kg (MTD=2.5 mg/kg) once on Day 1 of every 3 weeks (21-day cycle).
  HX008 will be administrated via intravenous infusion at 3 mg/kg once on Day 1 of every 3 weeks (21-day cycle).
  Interventions: Drug: MRG003+HX008

INTERVENTIONS:
Drug: MRG003+HX008 — Administered intravenously

SUMMARY:
The objective of this study is to assess the safety, efficacy, pharmacokinetics, and immunogenicity of MRG003 in combination with HX008 in patients with EGFR-positive advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
This study consists of two parts: Phase I and Phase II. The objective of this study is to assess the safety and tolerability of MRG003 in combination with HX008 in patients with EGFR-positive advanced or metastatic solid tumors; and to explore the maximum tolerated dose (MTD) and to determine the recommended phase II dose (RP2D) of combination therapy; and to evaluate the preliminary efficacy, pharmacokinetics, and immunogenicity of combination therapy in the targeted study population.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign the informed consent form and follow the requirements specified in the protocol.
2. Aged 18 to 75 (including 18 and 75), both genders.
3. BMI ≥17
4. Life expectancy ≥ 12 weeks.
5. Patients with EGFR-positive advanced or metastatic solid tumors, including non-small cell lung cancer (NSCLC), squamous cell carcinoma of head and neck (SCCHN), and nasopharyngeal carcinoma (NPC).
6. EGFR-positive determined by immunohistochemistry (except NSCLC, SCCHN and NPC).
7. Patients must have measurable lesions according to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
8. The score of ECOG for performance status is 0 or 1.
9. No severe cardiac dysfunction.
10. Acceptable liver, renal, and hematologic function.
11. Patients with childbearing potential must use effective contraception during the treatment and for 6 months after the last dose of treatment.

Exclusion Criteria:

1. History of hypersensitivity to any component of the investigational product.
2. Prior treatment with chemotherapy, biological therapy, immunotherapy, radiotherapy, investigational drugs, attenuated live vaccines, immunomodulators, CYP3A4 inhibitors/inducers, antibody-drug conjugates, Received major surgery without complete recovery, etc.
3. Treatment with MMAE/MMAF ADC drugs
4. Central nervous system metastasis.
5. Toxic reaction or abnormal value of laboratory test caused by previous anti-tumor treatment ≥ 2 (CTCAE v5.0)
6. Presence of peripheral neuropathy ≥ Grade 2.
7. Liver function Child Pugh Grade B or Grade C。
8. Pleural and peritoneal effusion or pericardial effusion with clinical symptoms requiring drainage.
9. Poorly controlled systemic diseases (hypertension and hyperglycemia, etc.)
10. Evidence of active infection of hepatitis B, hepatitis C or HIV.
11. Patients with poorly controlled heart diseases
12. History of ophthalmic abnormalities.
13. History of severe skin disease requiring oral or intravenous therapy.
14. History of interstitial pneumonia, radiation pneumonia, severe chronic obstructive pulmonary disease, severe pulmonary insufficiency, symptomatic bronchospasm, etc.
15. Active, known or suspected autoimmune disease or drug related immune disease or the disease history within the past 2 years.
16. The patient is using immunosuppressant or systemic hormone therapy.
17. Patients with any past arteriovenous bleeding within 3 months or current history of coagulation disorder.
18. Any clinically significant VTE occurred within 6 months.
19. Received allogeneic tissue/solid organ transplantation.
20. Inoculate live vaccine within 30 days before the first dose.
21. Patients with a positive serum pregnancy test or who are breast-feeding or who do not agree to take adequate contraceptive measures during the treatment and for 180 days after the last dose of study treatment.
22. History of other primary malignant tumor diseases.
23. Investigator considers which not suitable to participate in the clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Within 21 days after the first dose of the last patient of the MTD group
  MTD is the highest dose with the proportion of DLT less than 1/3
Recommended Phase II Dose (RP2D) | Baseline to study completion (up to 12 months)
  The dose level of MRG003 recommended for further clinical studies based on assessment of the safety, efficacy and PK data from this study.
Objective Response Rate (ORR) | Baseline to study completion (up to 12 months)
  ORR is defined as the proportions of patients with a complete response (CR) and partial response (PR). ORR will be assessed by investigator according to RECIST v1.1.

SECONDARY OUTCOMES:
Duration of Response (DOR) | Baseline to study completion (up to 12 months)
  DOR is defined as the duration from the initial recording of objective disease response to the first onset of tumor progression, or death of any cause.
Disease Control Rate (DCR) | Baseline to study completion (up to 12 months)
  DCR is defined as the proportion of subjects achieving CR, PR, and SD after treatment.
Progression Free Survival (PFS) | Baseline to study completion (up to 12 months)
  PFS is defined as the duration from the start of treatment to the onset of tumor progression or death of any cause.
Overall Survival (OS) | Baseline to study completion (up to 12 months)
  OS is defined as the duration from the start of treatment to death of any cause.
Immunogenicity (ADA) | Baseline to 90 days after the last dose.
  The proportion of patients with positive ADA results.
Adverse Events (AEs) | Baseline to 30 days after the last dose of study treatment
  Any reaction, side effect, or untoward event that occurs during the course of the clinical trial whether or not the event is considered related to the study drug.
Serious Adverse Events (SAEs) | Baseline to 90 days after the last dose of study treatment
  Adverse events that are difficult to deal with in clinical drug research
PK parameters: concentration-time curve | Baseline to 90 days after the last dose.
  Plot of drug concentration changing with time after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, M.D., Principal Investigator — Sun Yat-sen University
Locations (2):
- China (2):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Hunan Cancer Hospital, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No